CLINICAL TRIAL: NCT04611139
Title: Pilot Feasibility and Efficacy Trial of a Novel Reversible LSD1 Inhibitor SP-2577 (Seclidemstat) Plus Pembrolizumab in Select SWI/SNF-mutant Gynecologic Cancers
Brief Title: Pilot Trial of SP-2577 Plus Pembrolizumab in Select Gynecologic Cancers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Salarius discontinued support
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Salarius Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRI-SP-2577-001
Record Dates: First submitted 2020-09-24; First posted 2020-11-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: SCCOHT; Ovarian Clear Cell Tumor; Ovarian Endometrioid Adenocarcinoma; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SP-2577 Plus Pembrolizumab (Experimental)
  Interventions: Drug: SP-2577; Drug: Pembrolizumab

INTERVENTIONS:
Drug: SP-2577 — Daily oral doses
Drug: Pembrolizumab — 200mg Q3W by IV infusion

SUMMARY:
Open-label study of SF-2577 plus pembrolizumab in advanced, recurrent small cell ovarian cancer as well as select additional ovarian and endometrial cancers within the SWI/SNF pathway.

DETAILED DESCRIPTION:
This study is an open-label, non-randomized dose escalation and expansion study of the LSD inhibitor SP-2577 in combination with the anti PD- 1 antibody pembrolizumab in patients with advanced, recurrent small cell ovarian cancer of the hypercalcemic type (SCCOHT) as well as select additional ovarian and endometrial cancers with mutations in the genes within the SWI/SNF pathway (Ovarian Clear Cell Cancers (OCCC), Endometrioid Ovarian Cancers (EOC) and Endometrioid Endometrial Cancers (EEC).

ELIGIBILITY:
Inclusion Criteria:

* Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of small cell carcinoma of the ovary of hypercalcemic type (SCCOHT), ovarian clear cell carcinoma (OCCC), endometrioid ovarian carcinoma (EOC) or endometrioid endometrial carcinoma (EEC) with confirmed mutations in one of the SWI/SNF genes (SMARCA4, ARID1A) will be enrolled in this study.
* Patients must have received at least one prior regimen in the recurrent or advanced setting and must not be a candidate for other potentially curative treatment options.
* Not pregnant, breastfeeding and agrees to use contraceptive methods if child-bearing
* Provides written informed consent
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have provided archival tumor tissue sample or a newly obtained core or excisional biopsy of a tumor lesion not irradiated.
* ECOG of 0 to 1
* Adequate organ function

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation.
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent is allowed as long as patient did not have a serious (≥ Grade 3) immune related AE requiring treatment discontinuation or treatment with systemic steroids.
* Has received prior therapy with LSD1 targeted agents including monoamine oxidases for cancer therapy.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 half-lives whichever is shorter prior to the first dose of study treatment.
* Has received prior radiotherapy within 2 weeks of start of study treatment.
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has known active CNS metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of HIV, Hepatitis B, or known active Hepatitis C
* Has a known history of active TB
* Has clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality
* Is currently receiving any of the following substances and cannot be discontinued 14 days, or 5 half-lives for CYP inhibitors (whichever is shorter) prior to Cycle 1 Day 1
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Type of cancer being evaluated (ovarian and endometrial)
Enrollment: 0 (Actual)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incident of AEs | First dose to 90 days after last dose
  Incidence of Adverse Events (AEs) as measured by NCI CTCAE version 5.0
Incident of DLTs | First dose to 90 days after last dose
  Incidence of dose-limiting toxicities (DLTs) during the dose escalation phase
Overall Response Rate | Study enrollment until participant discontinuation, occurrence of PD or death (approximately 6 months to 3 years)
  Percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR), as determined by Investigator according to Response Evaluation in Solid Tumors (RECIST) v 1.1
Disease Control Rate | Study enrollment until PD or loss of clinical benefit (approximately 6 months to 3 years)
  Percentage of participants with Disease Control (complete response, partial response, or stable disease) as determined by RECIST v1.1
Duration of Response | Date of first occurrence of objective response to first documentation of PD (approximately 6 months to 3 years)
  Duration of Response as determined by the Investigator according to RECIST v1.1
Duration of Stable Disease | Date of first occurrence of stable disease to first documentation of PD (approximately 6 months to 3 years)
  Duration of Stable Disease as determined by the investigator according to RECIST v 1.1
Progression Free Survival | Start of treatment to first occurrence of PD or death (approximately 6 months to 3 years)
  Progression Free Survival (PFS) as determined by the Investigator according to RECIST v1.1
Overall Survival | Start of treatment to death (approximately 2 to 3 years)
  Overall Survival (OS) as determined by the Investigator according to RECIST v1.1

SECONDARY OUTCOMES:
Plasma Concentration of SP-2577 | 2 months
  Plasma concentration of seclidemstat (SP-2577)
ctDNA in blood and other body fluids | 6 months to 2 years
  Proportion of circulating tumor DNA ( ctDNA) in peripheral blood and other body fluids e.g. ascitic fluid
Target Inhibition in Tumor Biopsies | 6 months to 2 years
  Percentage of target inhibition by seclidemstat and pembrolizumab in tumor tissue biopsy specimens

CONTACTS AND LOCATIONS:
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No